CLINICAL TRIAL: NCT05783453
Title: CLINICAL EFFICACY OF EMOLLIENTS IN ATOPIC DERMATITIS PATIENTS: REDUCTION OF CRISES AND MAINTENANCE OF TREATMENT. STUDY UNDER NORMAL CONDITIONS OF USE AND DERMATOLOGICAL SUPERVISION
Brief Title: CLINICAL EFFICACY OF EMOLLIENTS IN ATOPIC DERMATITIS PATIENTS
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: 2122CBCL002
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis, eczema, emollient
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Emollients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cosmetic study — LIPIKAR BAUME LIGHT AP+M
  * Formula: 2039055 06
  * Aspect: Emulsion
  * Batch nº: RAUO0063
  * Expiry date: 10/2022
  * Application area: Face and Body
  * Application mode: Apply to face and body twice a day.
  * Quantity of product to be applied: About 1 flask (400g) per month
  Other Names: Emollient

SUMMARY:
his was a monocentric, intra-individual study, that was performed in at least 45 valid cases (50% children ≥3 YO; 50% adults). Study duration was 168 days with five (5) visits (D0, D14, D28, D84 and D168) to the research center.

Primary objective

* Evaluation of the efficacy of LIPIKAR BAUME LIGHT AP+M in decrease the SCORAD in child and adult subjects with mild atopic dermatitis after 14 and 28 days under normal conditions of use;
* Evaluation of the efficacy of LIPIKAR BAUME LIGHT AP+M in maintenance the SCORAD value in child and adult subjects with mild atopic dermatitis after 84 and 168 days under normal conditions of use.

Secondary objective

* Evaluation of flares quantity and severity during 84 and 168 days of use;
* Clinical evaluation of the improvement of skin parameters such as erythema, oedema, oozing, excoriation, lichenification, dryness and desquamation of a lesional and non-lesional skin from the same individual site by dermatologist after 14, 28, 84 and 168 days;
* Self-assessment of the improvement of skin parameters such as itching, tingling, burning by subjects after 14, 28, 84 and 168 days;
* Evaluate the perceived efficacy, cosmeticity and acceptability through a subjective evaluation questionnaire after 14, 28, 84 and 168 days;
* Evaluation of the improvement in skin barrier function by the loss of transepidermic water through instrumental measurements with the Tewameter® equipment on AF and UAF after 14, 28, 84 and 168 days;
* Evaluation of the improvement of skin moisturizing through instrumental measurements with Corneometer® equipment on AF and UAF after 14, 28, 84 and 168 days;
* The folliculitis incidence after 14, 28, 84 and 168 days;
* Assessment of the improvement of the impact of quality of life through a DLQI (Dermatology Life Quality Index) questionnaire after 14, 28, 84 and 168 days;
* Assessment of global tolerance through clinical dermatological evaluation and reports performed by the subjects after using the product after 14, 28, 84 and 168 days.
* Evaluation of total body skin dryness improvement after 14, 28, 84 and 168 days.
* Illustrative clinical pictures of one or two affected areas.

ELIGIBILITY:
Inclusion Criteria:

* Women or men, from 3 years old, being 50% children (≥3 years old ≤ 11 years and 11 months) and 50% adults;
* All phototypes (a good balance between the phototypes is not mandatory, but all phototypes should be included);
* Diagnosis of atopic dermatitis must meet Hanifin's criteria (at least 3 basic features and at least 3 minor features);
* Subject with mild atopic dermatitis present for at least 6 months before inclusion (SCORAD at inclusion < 25);
* Subjects that have an unchanged AD routine for at least 3 months, including to systematic use of topical or systemic antihistamines, topical or systemic corticoid, cyclosporin A and other immunosuppressant.
* Subject able to use the study product at least once a day during all study.
* Subject agreeing not to change their lifestyle during the study period (overbathing, being exposed to intense stress as change job, do a fast diet to loose weight…);
* Subject agreeing to use only the study product and no other topical treatment for the duration of the study (usual topical or oral treatment for AD is allowed);
* Subject capable of reading the documents presented to them, of adhering to the study regulations and accepting the limitations;
* Subject available to follow the study;
* Subject agreeing to participate and having signed the informed consent;
* Subject available to be contacted by phone throughout the study.

Exclusion Criteria:

* Breastfeeding, pregnant;
* Subject presenting with another dermatological condition that could interfere with clinical evaluation;
* Subject presenting a previous history of allergy to cosmetic products;
* Subject having received any systemic treatment, including PUVA therapy for atopic dermatitis in the month prior to Day 0;
* Subject having received phototherapy within 2 weeks before the first visit;
* Subject who intend to excessively expose themselves to the sun during the study;
* Subject known allergy to any component of the tested product (subjects will be asked if they have allergies to any ingredients and will be checked in the list if it is contained in the IP);
* Subject who have used any experimental treatment within 2 weeks before the first visit;
* Subject not presenting with the conditions needed to comply with the protocol;
* Subject unable to give their informed consent;
* Subject not available to follow the study in its entirety.

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: children and adult subjects with mild atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Improvement of SCORAD Score | baseline
  Decrease of SCORAD in child and adult subjects with mild atopic dermatitis after 14 and 28 days under normal conditions of use
Improvement of SCORAD Score | Day 14
  Decrease of SCORAD in child and adult subjects with mild atopic dermatitis after 14 and 28 days under normal conditions of use
Improvement of SCORAD Score | Day 28
  Decrease of SCORAD in child and adult subjects with mild atopic dermatitis after 14 and 28 days under normal conditions of use
Improvement of SCORAD Score | Day 84
  Maintenance of SCORAD in child and adult subjects with mild atopic dermatitis after 14 and 28 days under normal conditions of use
Improvement of SCORAD Score | Day 168
  Maintenance of SCORAD in child and adult subjects with mild atopic dermatitis after 14 and 28 days under normal conditions of use

SECONDARY OUTCOMES:
Flares | Baseline
  Evaluation of flares quantity and severity on a scale 0=none to 4=severe
Flares | Day 84
  Evaluation of flares quantity and severity on a scale 0=none to 4=severe
Flares | Day 168
  Evaluation of flares quantity and severity on a scale 0=none to 4=severe
Skin parameters | Baseline
  Improvement on a scale 0=none to 4=severe
Skin parameters | Day 14
  Improvement on a scale 0=none to 4=severe
Skin parameters | Day 28
  Improvement on a scale 0=none to 4=severe
Skin parameters | Day 84
  Improvement on a scale 0=none to 4=severe
Skin parameters | Day 156
  Improvement ona scale0=none to 4=severe
Product acceptability | Day 14
  Subject questionnaire
Product acceptability | Day 28
  Subject questionnaire
Product acceptability | Day 84
  Subject questionnaire
Product acceptability | Day 156
  Subject questionnaire
Skin hydration | Baseline
  Transepidermal water loss using tewameter
Skin hydration | Day 14
  Transepidermal water loss using tewameter
Skin hydration | Day 28
  Transepidermal water loss using tewameter
Skin hydration | Day 84
  Transepidermal water loss using tewameter
Skin hydration | Day 156
  Transepidermal water loss using tewameter
Skin moisturizing | Baseline
  Moisturising effect using corneometer
Skin moisturizing | Day 14
  Moisturising effect using corneometer
Skin moisturizing | Day 28
  Moisturising effect using corneometer
Skin moisturizing | Day 84
  Moisturising effect using corneometer
Skin moisturizing | Day 156
  Moisturising effect using corneometer
Folliculitis | Baseline
  scale 0=none to 4=severe
Folliculitis | Day 14
  scale 0=none to 4=severe
Folliculitis | Day 28
  scale 0=none to 4=severe
Folliculitis | Day 84
  scale 0=none to 4=severe
Folliculitis | Day 156
  scale 0=none to 4=severe
Evolution of Quality of life over time | Baseline
  DLQI (Dermatology Life Quality Index) questionnaire
Evolution of Quality of life over time | Day 14
  DLQI (Dermatology Life Quality Index) questionnaire
Evolution of Quality of life over time | Day 28
  DLQI (Dermatology Life Quality Index) questionnaire
Evolution of Quality of life over time | Day 84
  DLQI (Dermatology Life Quality Index) questionnaire
Evolution of Quality of life over time | Day 156
  DLQI (Dermatology Life Quality Index) questionnaire
local tolerance reporting | Day 14
  reporting of events
local tolerance reporting | Day 28
  reporting of events
local tolerance reporting | Day 84
  reporting of events
local tolerance reporting | Day 156
  reporting of events
Total body dryness | Baseline
  scale
Total body dryness | Day 14
  scale
Total body dryness | Day 28
  scale
Total body dryness | Day 84
  scale
Total body dryness | Day 156
  scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Miranda, MD, Study Director — CIDP Brasil
Locations (1):
- CIDP, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cestari S, Correia P, Kerob D. Emollients "Plus" are Beneficial in Both the Short and Long Term in Mild Atopic Dermatitis. Clin Cosmet Investig Dermatol. 2023 Aug 8;16:2093-2102. doi: 10.2147/CCID.S417622. eCollection 2023. PMID 37575149